CLINICAL TRIAL: NCT02601742
Title: Effectiveness of Oral Rehydration Therapy Supplemented With Zinc in the Management of Diarrhea Acute in Mexican Children: Randomized Double-blind Study
Brief Title: Effectiveness of Oral Rehydration Therapy Supplemented With Zinc in the Management of Diarrhea Acute
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Naval de Alta Especialidad - Escuela Medico Naval (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HGNAE-09
Record Dates: First submitted 2015-11-09; First posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-10

CONDITIONS: Diarrhea; Children
Keywords: zinc; Duration
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zinc group (Active Comparator): Pedialyte diarrhea oral electrolyte solution, 330 ml per day for 7 days
  Interventions: Other: Zinc group
- Placebo group (Placebo Comparator): Pedialyte oral electrolyte solution, 330 ml per day for 7 days
  Interventions: Other: Placebo group

INTERVENTIONS:
Other: Zinc group — Pedialyte diarrhea oral electrolyte solution, 330 ml per day for 7 days
  Other Names: Pedialyte diarrhea 45
  Arms: Zinc group
Other: Placebo group — Pedialyte oral electrolyte solution, 330 ml per day for 7 days
  Other Names: Pedialyte SR 45
  Arms: Placebo group

SUMMARY:
Acute diarrhea is the third cause of infant mortality in the world causing 15% of all deaths in children under 5 years and is responsible for nearly 1.4 million deaths in developing countries. It is considered a self-limiting disease and to this problem the recommendation of the World Health Organization (WHO) is the administration of zinc with low osmolarity oral dehydration salts for a period of 10-14 days which reduces the severity of the episode.

In Mexico COFEPRIS believes the zinc salt as a food supplement and not a drug and the above problem is presented in terms of prescribing and access of this salt to the general population. In Mexico the investigators have the provision and accessibility of low osmolarity oral dehydration salts supplemented with adequate doses of zinc, which is inexpensive for the general population and offering a solution in terms of supply and management.

The purpose of the study involves the evaluation Pedialyte diarrhea in the treatment of acute diarrhea in children under 5 years. The investigator sconsider the use of Pedialyte diarrhea eases their access to the population in general and it is low cost compared with the zinc salt that is sold only in specialized pharmacies under strict medical prescription Objective: Compare the duration of symptoms of acute diarrhea in the treatment with low osmolarity oral rehydration salts (Pedialyte) vs treatment of low osmolarity oral rehydration supplemented with zinc (Pedialyte diarrhea) Study Desing: Double blind, randomized, controlled.

DETAILED DESCRIPTION:
It will be conducted a randomized controlled double-blind in the Emergency service of the Naval General Hospital of High Specialty in the Mexico City. The period of patient inclusion in the study is October 2015 to November 2016.

The patients selections is the children between 6 months and 5 years who come to the emergency room with symptoms of acute diarrhea with up to 48 hours of starting the disease, it will proceed to questioning and to assess vital signs and thorough physical examination for determine the degree of dehydration, nutritional status and rule out diagnosis of abdominal pathology emergency.

Selection criteria Inclusion

* Patients 6 months to 5 years old with acute diarrhea
* Patients in their first 48 hours of onset diarrhea
* Dehydration mild to moderate according to WHO clinical scale
* Both sexes
* Outpatients

Exclusion

* Patients with vomit (10 or more)
* Hemodynamic Instability
* Dehydration severe
* Patients with heart disease
* Patients with a history of prematurity.
* Patients with chronic diarrhea
* Patients whose parents refuse to provide written informed consent
* Patients who do not comply with treatment correctly
* Patients with suspected surgical pathology

Elimination

* Patients with severe dehydration
* Patients in whom the parents decline for informed consent

ELIGIBILITY:
Inclusion Criteria:

* Patients 6 months to 5 years old with acute diarrhea
* Patients in their first 48 hours of onset diarrhea
* Dehydration mild to moderate according to WHO clinical scale
* Both sexes
* Outpatients

Exclusion Criteria:

* Patients with vomit (10 or more)
* Hemodynamic Instability
* Severe dehydration
* Patients with heart disease
* Patients with a history of prematurity.
* Patients with chronic diarrhea
* Patients whose parents refuse to provide written informed consent
* Patients who do not comply with treatment correctly
* Patients with suspected surgical pathology

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-01 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Number of bowel movements per day | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: María del Carmen Yebra Cano, Medicina, Principal Investigator — Secretaria de Marina-Armada de México (Mexican Navy)

REFERENCES:
- [Background] Liu L, Johnson HL, Cousens S, Perin J, Scott S, Lawn JE, Rudan I, Campbell H, Cibulskis R, Li M, Mathers C, Black RE; Child Health Epidemiology Reference Group of WHO and UNICEF. Global, regional, and national causes of child mortality: an updated systematic analysis for 2010 with time trends since 2000. Lancet. 2012 Jun 9;379(9832):2151-61. doi: 10.1016/S0140-6736(12)60560-1. Epub 2012 May 11. PMID 22579125
- [Background] Gupta GR. Tackling pneumonia and diarrhoea: the deadliest diseases for the world's poorest children. Lancet. 2012 Jun 9;379(9832):2123-4. doi: 10.1016/S0140-6736(12)60907-6. No abstract available. PMID 22682449
- [Background] Aurelio Mejia y cosl., Analisis de costo beneficio de la suplementación con Zinc en el tratamiento de la diarrea aguda en niños menores de 5 años en Colombia, publicado en ESPGHAN 2015
- [Background] Scrimgeour, A.; Condlin, M.; Otieno, L.; Bovill, M. Zinc intervention strategies: Costs and health benefits. In Nutrients, Dietary Supplements, and Nutriceuticals; Gerald, J.K., Watson, R.R., Preedy, V.R., Eds.; Humana Press: 201
- [Background] WHO/UNICEF. Joint Statement on the Clinical Management of Acute Diarrhoea; UNICEF: 2004
- [Background] Benguigui Y, Bernal C, Figueroa D, eds. Manual de Tratamiento de la Diarrea en Nin˜os. Washington, DC: Panamerican Health Organization/ Organización Panamericana de la Salud; 2008
- [Background] Malek MA, Curns AT, Holman RC, Fischer TK, Bresee JS, Glass RI, Steiner CA, Parashar UD. Diarrhea- and rotavirus-associated hospitalizations among children less than 5 years of age: United States, 1997 and 2000. Pediatrics. 2006 Jun;117(6):1887-92. doi: 10.1542/peds.2005-2351. PMID 16740827
- [Background] Majowicz SE, McNab WB, Sockett P, Henson TS, Dore K, Edge VL, Buffett MC, Fazil A, Read S, McEwen S, Stacey D, Wilson JB. Burden and cost of gastroenteritis in a Canadian community. J Food Prot. 2006 Mar;69(3):651-9. doi: 10.4315/0362-028x-69.3.651. PMID 16541699
- [Background] Lazzerini M, Ronfani L. Oral zinc for treating diarrhoea in children. Cochrane Database Syst Rev. 2012 Jun 13;(6):CD005436. doi: 10.1002/14651858.CD005436.pub3. PMID 22696352
- [Background] Liberato SC, Singh G, Mulholland K. Zinc supplementation in young children: A review of the literature focusing on diarrhoea prevention and treatment. Clin Nutr. 2015 Apr;34(2):181-8. doi: 10.1016/j.clnu.2014.08.002. Epub 2014 Aug 13. PMID 25176404
- [Background] Dr Rul L. Riveron Corteguera, Fisiopatología de la diarrea aguda, Hospital pediátrico docente de la Habana 2009
- [Background] King JC, Shames DM, Woodhouse LR. Zinc homeostasis in humans. J Nutr. 2000 May;130(5S Suppl):1360S-6S. doi: 10.1093/jn/130.5.1360S. PMID 10801944
- [Background] Baqui AH, Black RE, El Arifeen S, Yunus M, Chakraborty J, Ahmed S, Vaughan JP. Effect of zinc supplementation started during diarrhoea on morbidity and mortality in Bangladeshi children: community randomised trial. BMJ. 2002 Nov 9;325(7372):1059. doi: 10.1136/bmj.325.7372.1059. PMID 12424162
- [Background] Fischer Walker CL, Fontaine O, Young MW, Black RE. Zinc and low osmolarity oral rehydration salts for diarrhoea: a renewed call to action. Bull World Health Organ. 2009 Oct;87(10):780-6. doi: 10.2471/blt.08.058990. PMID 19876545
- [Background] Maggini S, Wenzlaff S, Hornig D. Essential role of vitamin C and zinc in child immunity and health. J Int Med Res. 2010 Mar-Apr;38(2):386-414. doi: 10.1177/147323001003800203. PMID 20515554
- See also: Encuesta Nacional de Salud y Nutrición 2012 — http://www.insp.mx